CLINICAL TRIAL: NCT05446896
Title: Setting-up Of A Mechanical Ventilator With An Augmented Reality Guide: A Prospective, Randomized Pilot Trial
Brief Title: Effectiveness of AR in Ventilator Setting Education.
Acronym: AR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Meong Hi Son, department of Pediatrics, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-12-112-001
Record Dates: First submitted 2022-06-25; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: Nursing Education
Keywords: Ventilator, Nursing, Education, Augmented reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR group (Experimental): participants in the AR group were guided by AR-based instructions and requested assistance with the head-mounted device.
  Interventions: Device: AR guidance with Hololens 2
- manual group (No Intervention): Participants in the manual group used a printed manual and made a phone call for assistance.

INTERVENTIONS:
Device: AR guidance with Hololens 2 — The AR instructions were developed as a step-by-step guide with the same text and images as in the printed manual, utilizing the dynamic 365 Guide (Software, Microsoft Corporation, Redmond, WA, USA). The AR instructions were delivered using the Microsoft HoloLens 2.
  Arms: AR group

SUMMARY:
This study aimed to determine the feasibility and effectiveness of an augmented reality (AR)-based self-learning platform for novices to set up a ventilator without on-site assistance. This was a prospective randomized controlled pilot study conducted at Samsung Medical Center, Korea from January to February 2022. Nurses with no prior experience of MV or AR were enrolled. We randomized the participants into two groups: manual and AR groups. Participants in the manual group used a printed manual and made a phone call for assistance, whereas participants in the AR group were guided by AR-based instructions and requested assistance with the head-mounted device (HMD). We compared the overall score of the procedure, required level of assistance, and user's experience between the groups.

DETAILED DESCRIPTION:
Background: Recently, the demand for mechanical ventilation (MV) has increased with the COVID-19 pandemic; however, the conventional approaches to MV training are resource-intensive and require on-site training. Consequently, the need for independent learning platforms with remote assistance in institutions without resources has surged.

Objective:

This study aimed to determine the feasibility and effectiveness of an augmented reality (AR)-based self-learning platform for novices to set up a ventilator without on-site assistance.

Method:

This was a prospective randomized controlled pilot study conducted at Samsung Medical Center, Korea from January to February 2022. Nurses with no prior experience of MV or AR were enrolled. We randomized the participants into two groups: manual and AR groups. Participants in the manual group used a printed manual and made a phone call for assistance, whereas participants in the AR group were guided by AR-based instructions and requested assistance with the head-mounted device (HMD). We compared the overall score of the procedure, required level of assistance, and user's experience between the groups.

ELIGIBILITY:
Inclusion Criteria:

We enrolled nurses who had no prior experience with ventilator setup or AR systems, regardless of their work department or age.

Exclusion Criteria:

We excluded nurses who had already experienced setting up a ventilator or who had trouble wearing or using a head-mounted device (HMD).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
the overall score of the procedure | 30 minutes
  a 100-point scale converted from the original score. The participants scored 1 point for each step if they successfully finished the step within five minutes and obtained a maximum score of 35.

SECONDARY OUTCOMES:
the required level of assistance | 30 minutes
  The number of steps needed assistance to complete the procedure

OTHER OUTCOMES:
Usability | 30 minutes
  System usability scale

CONTACTS AND LOCATIONS:
Overall Officials: Meong Hi Son, MD, Principal Investigator — Department of Pediatrics Samsung Medical Center and Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Centre, Seoul, South Korea

REFERENCES:
- [Derived] Heo S, Moon S, Kim M, Park M, Cha WC, Son MH. An Augmented Reality-Based Guide for Mechanical Ventilator Setup: Prospective Randomized Pilot Trial. JMIR Serious Games. 2022 Jul 22;10(3):e38433. doi: 10.2196/38433. PMID 35867382